CLINICAL TRIAL: NCT07264478
Title: Beijing Children's Hospital, Capital Medical University, China National Clinical Research Center of Respiratory Diseases, National Center for Children's Health, Beijing, China
Brief Title: Diagnosis and Treatment Status and Medical Burden of Respiratory Syncytial Virus Infection in Children in China
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, professor, Beijing Children's Hospital
Other Study IDs: BCH lung 22
Record Dates: First submitted 2023-10-12; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: RSV Infection; Disease Burden
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: uninvolved — uninvolved

SUMMARY:
To understand the diagnosis and treatment status and medical burden of respiratory syncytial virus (RSV) infection in children in China, and to provide scientific basis for formulating prevention and treatment strategies for children. According to the seven administrative regions of China, namely Northeast, North, Northwest, Southwest, Central, South and East China, 1-3 children's medical institutions were selected from each region, and the cases of bronchiolitis or pneumonia admitted to hospitals and diagnosed as RSV positive by etiology during January 1, 2017 to December 31, 2021 were selected. Demographic data and clinical information were collected, and subgroup analysis was designed to explore the relationship between them and medical expenses and clinical treatment burden.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients under 18 years of age with an etiological diagnosis of RSV-positive bronchiolitis or pneumonia

Exclusion Criteria:

Inpatients under 18 years of age with an etiological diagnosis of RSV-positive bronchiolitis or pneumonia are excluded from any of the following criteria:

1. Pneumonia occurring 48 hours after hospitalization;
2. Combined with bronchial foreign body;
3. Participants in clinical trials of drugs or medical devices;
4. Not complete personal and family history and other relevant information.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: According to the seven administrative regions of China, namely Northeast, North, Northwest, Southwest, Central, South and East China, 1-3 children's medical institutions were selected from each region, and the cases of bronchiolitis or pneumonia admitted to hospitals and diagnosed as RSV positive by etiology during January 1, 2017 to December 31, 2021 were selected. A total of 11 hospitals were selected, each with 100 children, a total of 1100 cases
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
hospitalization costs | duration of hospital stay
  hospitalization costs,pharmcost,testcost,testcost

SECONDARY OUTCOMES:
hospital day | duration of hospital stay
  duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No